CLINICAL TRIAL: NCT05857319
Title: Assessment of the Impact of Short, Medium and Long-term Weight Loss, Obtained by a Standardized Nutritional and Psycho-Behavioral Rehabilitation Program (RNPC Program) and in Real Life Conditions, in Obese or Overweight Patients
Brief Title: Study Consortium for Evaluation of RNPC Program in Obese and Overweight Patients (SCOOP-RNPC)
Acronym: SCOOP-RNPC
Status: Not yet recruiting | Type: Observational
Sponsor: Groupe Éthique et Santé (Industry)
Collaborators: University Grenoble Alps (Other); Novo Nordisk A/S (Industry); Lyon Est University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-A01599-34
Record Dates: First submitted 2023-03-29; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Overweight and Obesity; Cardiovascular Diseases; Metabolic Disease; Diabete Type 2; Sleep Apnea, Obstructive; NAFLD; NASH
Keywords: Prospective Interventional Study; Real-Life Conditions; RNPC Program
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases; Metabolic Diseases; Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- General Cohort: The General Cohort includes all participants of the study. These are enrolled in the RNPC Program and will provide clinical and biological data usually collected in the RNPC centers, enriched by data from additional clinical and biological examinations as well as by self-questionnaires completed by the participants.
- Connected Objects Group: Depending on the RNPC center in which the participant is followed, he/she will be offered to be part of the Connected Objects subgroup, with specific additional examinations on inclusion as well as at certain key times of the intervention:
  * Measurement of anthropometric parameters and evaluation of arterial stiffness using the Body Cardio connected scale (Withings).
  * Sleep evaluation using the Sleep Analyzer (Withings); Measurements taken at the participant's home.
  Interventions: Behavioral: Nutritional Psycho-Behavioral Reeducation Program
- Obstructive Sleep Apnea Syndrome (OSAS) Group: Depending on the RNPC center in which the participant is followed, he/she will be offered to be part of the OSAS subgroup, with specific additional examinations on inclusion as well as at certain key times of the intervention:
  * Sleep assessment and diagnosis of OSAS (if applicable) via the Sunrise device. Measurements taken at the participant's home.
  Interventions: Behavioral: Nutritional Psycho-Behavioral Reeducation Program
- Neuropathies Group: Depending on the RNPC center in which the participant is followed, he/she will be offered to be part of the Neuropathies subgroup, with specific additional examinations at each visit:
  * Detection of diabetic neuropathies using SUDOSCAN/EZSCAN technology (Withings). Measurements taken at the center.
  Interventions: Behavioral: Nutritional Psycho-Behavioral Reeducation Program

INTERVENTIONS:
Behavioral: Nutritional Psycho-Behavioral Reeducation Program — The RNPC Program is based on a clinical protocol in three successive phases:
  1. A weight loss phase during which food intake is restricted to 800-1000 kcal per day, with a nutrient distribution of 60% protein, 25% carbohydrates and 15% lipids. Patients eat two meals a day consisting of meat/fish/eggs/shellfish and vegetables, supplemented by products enriched in proteins, vitamins and minerals, and depleted in carbohydrates and lipids.
  2. A stabilization phase specifically established for each patient according to their weight loss and their daily caloric needs, allowing them to gradually return to a balanced diet, with a nutrient distribution of 25% protein, 45% carbohydrates and 30% lipids. During this phase, the consumption of meal supplements gradually decreases.
  3. A phase of return to dietary balance, unlimited in time, based on the precepts of the Mediterranean diet.
  Each patient is followed every 14 days by a dietitian during the entire program.
  Other Names: RNPC Program
  Groups: Connected Objects Group; Neuropathies Group; Obstructive Sleep Apnea Syndrome (OSAS) Group

SUMMARY:
The investigators hypothesize that weight loss obtained with the French RNPC weight reduction program is beneficial for the general health of overweight/obese patients in the medium term.

The objective of this cohort study is to demonstrate the effectiveness of the RNPC program on the reduction of drug or instrumental treatments (for example, continuous positive pressure ventilation for the treatment of sleep apnea syndrome) and the improvement of overweight/obesity-associated comorbidities in the medium term.

This is a multicenter clinical study, as part of routine care, with standardized nutritional care (RNPC Program) in all RNPC centers in France. A cohort will be formed based on the clinical and biological data usually collected in the centers, enriched by data from additional clinical and biological examinations as well as by self-questionnaires completed by the participants. About 10,000 overweight or obese participants will be included for 2 years and followed 5 years.

The SCOOP-RNPC study will have benefits for individual participants, for the scientific community in terms of knowledge acquired and for society with a better definition of the impact of treatments.

Responding to the major public health issue represented by overweight, this prospective cohort of overweight or obese patients will make it possible to evaluate, in real-life conditions, the effects of weight loss obtained by the RNPC Program in the short, medium and long term on biological parameters predictive of cardiometabolic risk, drug consumption, quality of life, diet and eating behavior, sleep, physical activity, stress/anxiety, as well as depression.

This cohort will make it possible to identify clinical phenotypes and biomarkers to optimize the personalization of the management of overweight or obese patients, in particular those at risk of developing comorbidities associated with excess weight.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than or equal to 25 kg/m² and/or waist circumference greater than or equal to 80 cm in women and 94 cm in men;
* Possessing a personal smartphone;
* Subjects subject to the French health system;
* Subjects able to sign the informed consent.

Exclusion Criteria:

* Persons refusing to sign the participation consent;
* Pregnant, parturient and breastfeeding women;
* Persons with missing limb(s);
* People with an electrical medical device such as a pacemaker, battery, insulin pump or cochlear implant;
* People carrying any metallic material present in the body, such as prostheses or screws;
* Persons under guardianship;
* Subject in period of exclusion from another study;
* Person deprived of liberty by judicial or administrative decision;
* Person subject to a legal protection measure, who cannot be included in clinical trials;
* People with an open wound or bleeding on the palms of the hands or soles of the feet (Neuropathy group only).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All new patients committing to follow the RNPC Program in the RNPC investigator centers are potentially eligible for the study and will be offered to participate.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2030-07-15 (Estimated); Study Completion 2030-07-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the national RNPC weight reduction program on the change of treatments (drug or instrumental treatments) or in the comorbidities of overweight/obesity. | Assessed at baseline, after the first phase of the intervention, after the second phase of the intervention, and every year after completion of the intervention for 5 years.
  The primary endpoint is defined as the number of participants who had at least one dose change of their initial drug and/or instrumental treatment(s) and/or disappearance of comorbidities of overweight/obesity (indicative list of comorbidities possibly concerned: arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, obstructive sleep apnea syndrome, depression, pain, etc.) at the end of the program (minimum duration of 6 months but not exceeding one year).

SECONDARY OUTCOMES:
Weight | Data collected through study completion for 5 years.
  Weight in kilograms (kg) of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Body mass index (BMI) | Data collected through study completion for 5 years.
  BMI, calculated according to the formula: [weight (in kg) ÷ height x height (in meters)], of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Waist circumference | Data collected through study completion for 5 years.
  Waist circumference (in centimeters) of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Hip circumference | Data collected through study completion for 5 years.
  Hip circumference (in centimeters) of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Waist-to-hip circumference ratio | Data collected through study completion for 5 years.
  Waist-to-hip circumference ratio of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Neck circumference | Data collected through study completion for 5 years.
  Neck circumference (in centimeters) of identified subgroups, defined according to the comorbidities initially present (i.e. before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Muscle mass percentage | Data collected through study completion for 5 years.
  Muscle mass percentage of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Fat mass percentage | Data collected through study completion for 5 years.
  Fat mass percentage of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Water mass percentage | Data collected through study completion for 5 years.
  Water mass percentage of identified subgroups, defined according to the comorbidities initially present (i.e., before the start of the intervention; arterial hypertension, glucose intolerance, type 2 diabetes, dyslipidemia, OSAS) and the level of initial BMI.
Percentage of participants who changed BMI category at the end of each phase of the RNPC program. | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  BMI category is determined at the initial visit, at the end of the weight loss phase and at the end of the stabilization phase.
  The following BMI categories will be considered: < 25 kg/m², ≥ 25 and < 30 kg/m², ≥ 30 and < 35 kg/m², ≥ 35 and < 40 kg/m², ≥ 40 kg/m².
Pain assessment | Data collected through study completion for 5 years.
  Pain will be assessed by the dietitian using a visual analogue scale (VAS), with a score from 0 to 10.
Fasting glycemia | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Fasting glycemia in g/L.
Fasting insulinemia | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Fasting insulinemia in mUI/L.
HbA1c percentage | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Hemoglobin A1c (HbA1c; glycated hemoglobin), only in participants with type 2 diabetes.
HOMA-IR index | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  HOMA-IR (homeostasis model assessment of insulin resistance) index is calculated according to the formula: [fasting insulinemia (microU/L) x fasting glycemia (nmol/L) / 22.5].
TyG index | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  TyG (triglyceride-glucose) index is calculated according to the formula: [ln (triglyceridemia in g/L) x (fasting glycemia in g/L) / 2].
QUICKI | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  QUICKI (quantitative insulin sensitivity check index) is calculated according to the formula: [1 / (log fasting insulinemia in mIU/L) + (log fasting glycemia in g/L)].
Level of total cholesterol | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of total cholesterol (in g/L) in blood samples.
Level of HDL-cholesterol | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of HDL-cholesterol (in g/L) in blood samples.
Level of LDL-cholesterol | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of LDL-cholesterol (in g/L) in blood samples.
Level of triglycerides | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of triglycerides (in g/L) in blood samples.
SCORE2/SCORE2-OP score | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Calculation of SCORE2 (or SCORE2-OP for people aged ≥ 70 years) score, for evaluation of the overall cardiovascular risk score over 10 years, is based on the following biological parameters:
  * Age (year);
  * Systolic blood pressure (mm Hg);
  * Level of total cholesterol (g/L);
  * Level of HDL-cholesterol (g/L);
  * Blood pressure medication (yes or no);
  * Cigarette smoker (yes or no);
  * Diabetes present or not.
Changes in the presence or not of a metabolic syndrome | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Criteria for metabolic syndrome were determined by the International Diabetes Federation in 2005:
  Waist circumference ≥ 94 cm (men) and ≥ 80 cm (women), plus at least 2 of the following criteria:
  * Fasting glycemia ≥ 1 g/L and/or diagnosis of diabetes and/or treatment for diabetes;
  * Level of HDL cholesterol < 0.4 g/L (men) and < 0.5 g/L (women) or specific treatment for this lipid disorder;
  * Triglyceridemia ≥ 1.5 g/L or specific treatment for this lipid disorder;
  * Blood pressure ≥ 130/85 mm Hg (≥ 130/80 mm Hg if diabetes) and/or treatment for high blood pressure.
Level of ALAT | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of ALAT (alanine aminotransferase; in UI/L) in blood samples.
Level of ASAT | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of ASAT (alanine aminotransferase) in blood samples.
Ferritinemia | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of ferritin (in ng/mL) in blood samples.
FibroMeter score | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Calculation of FibroMeter score is based on the following biological parameters:
  * Platelet count (G/L);
  * ALAT (UI/L);
  * ASAT (UI/L);
  * Fasting glycemia (g/L);
  * Ferritinemia.
Level of GGT | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of GGT (gamma-glutamyl transferase; in g/L) in blood samples.
Creatininemia | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Creatininemia in mg/L.
Creatininuria | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Creatininuria (in mg/L), dosed on a single sample of urine from the first urination in the morning.
Microalbuminuria | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Microalbuminuria (in mg/L), dosed on a single sample of urine from the first urination in the morning.
MDRD score | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  MDRD (modification of diet in renal disease) score is calculated according to the formula: [186 x (creatininemia in mg/L/88.4) x (Age) x (0.742 if female) x (1.210 if black)].
Albumin-creatinine ratio | Assessed at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Urinary albumin-creatinine ratio.
Levels of plasma amino acids (glutamine, glutamate and alanine) | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of Plasma amino acids (glutamine, glutamate and alanine; in µmol/L). Intestinal and hepatic gluconeogenesis will be evaluated by quantitative determination of plasma amino acids (glutamine, glutamate and alanine), associated with the determination of lactate, pyruvate, glycerol and fatty acid levels.
Level of lactate | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of lactate (in mg/L) in blood samples. Intestinal and hepatic gluconeogenesis will be evaluated by quantitative determination of plasma amino acids (glutamine, glutamate and alanine), associated with the determination of lactate, pyruvate, glycerol and fatty acid levels.
Level of pyruvate | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of pyruvate (in mg/L) in blood samples. Intestinal and hepatic gluconeogenesis will be evaluated by quantitative determination of plasma amino acids (glutamine, glutamate and alanine), associated with the determination of lactate, pyruvate, glycerol and fatty acid levels.
Level of glycerol | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of glycerol (in mg/L) in blood samples. Intestinal and hepatic gluconeogenesis will be evaluated by quantitative determination of plasma amino acids (glutamine, glutamate and alanine), associated with the determination of lactate, pyruvate, glycerol and fatty acid levels.
Level of fatty acids | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Dosage of fatty acids in blood samples. Intestinal and hepatic gluconeogenesis will be evaluated by quantitative determination of plasma amino acids (glutamine, glutamate and alanine), associated with the determination of lactate, pyruvate, glycerol and fatty acid levels.
Blood pressure | Data collected through study completion for 5 years.
  Measurement of systolic and diastolic blood pressure (in mm Hg).
Score to the Epworth Sleepiness Scale (ESS) questionnaire | Questionnaire completed at baseline, after the first phase of the intervention, after the second phase of the intervention, and every year after completion of the intervention for 5 years.
  Score calculated from participants' responses to the sleep-related self-administered questionnaire Epworth Sleepiness Scale (ESS), completed online, between two visits to the RNPC center.
Score to the Pittsburgh Sleep Quality Index (PSQI) questionnaire | Questionnaire completed at baseline, after the first phase of the intervention, after the second phase of the intervention, and every year after completion of the intervention for 5 years.
  Score calculated from participants' responses to the sleep-related self-administered questionnaire Pittsburgh Sleep Quality Index (PSQI), completed online, between two visits to the RNPC center.
Score to the Insomnia Severity Index (ISI) questionnaire | Questionnaire completed at baseline, after the first phase of the intervention, after the second phase of the intervention, and every year after completion of the intervention for 5 years.
  Score calculated from participants' responses to the sleep-related self-administered questionnaire Insomnia Severity Index (ISI), completed online, between two visits to the RNPC center.
Score to the Chronotype questionnaire | Questionnaire completed at baseline.
  Score calculated from participants' responses to the self-administered Chronotype questionnaire, completed online, between two visits to the RNPC center.
Evolution of Obstructive Sleep Apnea Syndrome (OSAS) | Data collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  OSAS is defined according to the apnea-hypopnea index (AHI), collected by connected devices (Sleep Analyzer and Sunrise). Only participants in the Connected Objects group and in the OSAS group will be concerned.
Score to the 5-level EQ-5D version (EQ-5D-5L) questionnaire | Questionnaire completed at baseline, after the first phase of the intervention, after the second phase of the intervention, and every year after completion of the intervention for 5 years.
  Score calculated from participants' responses to the quality-of-life EQ-5D version (EQ-5D-5L) self-administered questionnaire, completed online, between two visits to the RNPC center.
Score to the EQVOD ('Échelle de Qualité de Vie, Obésité et Diététique') French questionnaire | Questionnaire completed at baseline, after the first phase of the intervention, after the second phase of the intervention, and every year after completion of the intervention for 5 years.
  Score calculated from participants' responses to the quality-of-life EQVOD French self-administered questionnaire, completed online, between two visits to the RNPC center.
Score to the Food Frequency Questionnaire (FFQ) | Questionnaire completed at baseline.
  Score calculated from participants' responses to the eating habits-related Food Frequency Questionnaire (FFQ) self-administered questionnaire, completed online, between two visits to the RNPC center.
Score to the Three-Factor Eating Questionnaire (TFEQ) | Questionnaire completed collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Score calculated from participants' responses to the eating behavior-related Three-Factor Eating Questionnaire (TFEQ) self-administered questionnaire, completed online, between two visits to the RNPC center.
Score to the Hospital Anxiety and Depression (HAD) scale | Questionnaire completed collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Score calculated from participants' responses to the stress, anxiety and depression-related Hospital Anxiety and Depression (HAD) scale, self-administered and completed online, between two visits to the RNPC center.
Score to the Perceived Stress Scale (PSS) | Questionnaire completed collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Score calculated from participants' responses to stress-related Perceived Stress Scale (PSS) self-administered questionnaire, completed online, between two visits to the RNPC center.
Responses to the general questionnaire | Questionnaire completed at baseline and every year after completion of the intervention for 5 years.
  Responses collected from a general questionnaire (information about socio-cultural level, life environment, family and social life, married life, etc.), completed online, between two visits to the RNPC center.
Arterial stiffness | Data collected at baseline, after having lost 10% of initial body weight, after the first phase of the intervention and after the second phase of the intervention, at least.
  Arterial stiffness will be assessed by measuring pulse wave velocity (PWV), data collected regularly by the Body Cardio connected scale. Only participants in the Connected Objects group will be concerned.
Prevalence of peripheral neuropathies at the start of the intervention | Data collected at baseline.
  The SUDOSCAN device provides results as conductances of the feet and hands (in microsiemens; with the average of the left and right sides). High conductance levels are correlated with normal sweat function and healthy innervation (small C-fibers). Low conductances represent peripheral autonomic neuropathy. The EZSCAN risk score (classified in quadrants: at risk/moderate/no risk, with a color code) determined from these measures indicates the risk of developing diabetes. Only participants in the Neuropathies group will be concerned.
Evolution of peripheral neuropathies | Data collected at baseline, after having lost 10% of initial body weight, after the first phase of the intervention and after the second phase of the intervention, at least.
  The SUDOSCAN device provides results as conductances of the feet and hands (in microsiemens; with the average of the left and right sides). High conductance levels are correlated with normal sweat function and healthy innervation (small C-fibers). Low conductances represent peripheral autonomic neuropathy. The EZSCAN risk score (classified in quadrants: at risk/moderate/no risk, with a color code) determined from these measures indicates the risk of developing diabetes. Only participants in the Neuropathies group will be concerned.
Score to the Baecke questionnaire | Questionnaire completed collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Score calculated from participants' responses to the physical-activity-related Baecke self-administered questionnaire, completed online between two visits to the RNPC center.
Distance traveled (by foot) per week | Data collected through study completion for 5 years.
  The dietician will collect, directly from the pedometer application of the participant's smartphone, the distance traveled by foot (in meters) of the past week.
Number of steps per week | Data collected through study completion for 5 years.
  The dietician will collect, directly from the pedometer application of the participant's smartphone, the number of steps of the past week.
Dropout rate | Assessed collected at baseline, after the first phase of the intervention and after the second phase of the intervention.
  Drop-out of participants (who stopped the weight loss program before the end of the stabilization phase) during the intervention in all subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, MD, PhD, Principal Investigator — Grenoble Alpes University, INSERM U1300; Arne Astrup, MD, PhD, Study Chair — Department of Obesity and Nutritional Sciences, Novo Nordisk Foundation; Gilles Mithieux, PhD, Study Chair — Lyon Est University, INSERM U1213

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fabre O, Bailly S, Mithieux G, Legrand R, Costentin C, Astrup A, Pepin JL. Long-term trajectories of weight loss and health outcomes: protocol of the SCOOP-RNPC nationwide observational study. BMJ Open. 2024 Jul 11;14(7):e082575. doi: 10.1136/bmjopen-2023-082575. PMID 38991672